CLINICAL TRIAL: NCT06828081
Title: Comparative Effects of Getting it Right AddressingShoulderPain(GRASP)Trial and Rotator Cuff Strengthening Exercise Program Among Military Sports for Rotator Cuff Tendinopathy
Brief Title: Comparative Effects of Getting it Right Addressing Shoulder Pain and Rotator Cuff Strengthening Exercise Military Sports
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0426
Record Dates: First submitted 2024-11-18; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Sports Physical Therapy
Keywords: Rotator cuff tendinopathy; GRASP trails; Military sports; Shoulder pain
MeSH Terms: conditions — Shoulder Pain | interventions — Range of Motion, Articular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Range of Motion Exercises (Experimental): Will get standard shoulder muscle exercises, including rigid and stretchy ones with bands that offer resistance.
  Interventions: Other: Range of Motion Exercises
- Strengthening exercises with theraband (Experimental): They will go through the GRASP method, which involves special workouts just for them, teaching them about their health and ways to deal with pain.
  Interventions: Other: Strengthening exercises with theraband

INTERVENTIONS:
Other: Range of Motion Exercises — Will get standard shoulder muscle exercises, including rigid and stretchy ones with bands that offer resistance.
  Arms: Range of Motion Exercises
Other: Strengthening exercises with theraband — They will go through the GRASP method, which involves special workouts just for them, teaching them about their health and ways to deal with pain.
  Arms: Strengthening exercises with theraband

SUMMARY:
This research will use a randomized clinical trial (RCT) method to get military athletes with rotator cuff tendinopathy. People will be chosen at random to either get the GRASP method or normal exercises for making the shoulder muscles stronger. The main things the investigator will look at are how bad the pain is how well the shoulder works and if they can go back to work or sports. Tests will be done at the start, right after a treatment, and later times to measure the short-term and long-term advantages of the treatments. This study's careful way of doing things aims to provide strong information for military sports medicine. It helps doctors in treating shoulder problems like rotator cuff tendinopathy.

DETAILED DESCRIPTION:
The rationale for conducting this study lies in the critical need to address rotator cuff tendinopathy, a prevalent and debilitating issue among military athletes. The unique demands placed on military personnel, involving repetitive overhead tasks and rigorous training, contribute significantly to the higher incidence of rotator cuff problems. The impact of this condition on performance, readiness, and overall well-being in the military cannot be overstated.

In the end, the plan for this study wants to fix a gap in what we know right now about dealing with muscle problems in military sports players' shoulders. This study looks at the GRASP trial methods and compares them with standard rotator cuff exercises. It aims to improve treatments and help military staff be healthier and work better.

ELIGIBILITY:
Inclusion Criteria:

* People in the military who are between 18 and 50 years old.
* Active participation in sports activities for the military.
* Diagnosing rotator cuff tendon pain in medical practice.
* Basic shoulder movement within a certain range of motion.

Exclusion Criteria:

* History of shoulder surgery.
* Systemic inflammatory diseases.
* Disorders of the brain or mind that affect physical actions.
* Not being able to stick to the plan for later.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | 5-6weeks
  The Western Ontario Rotator Cuff Index (WORC) is a self-reported questionnaire that evaluates the quality of life in individuals with rotator cuff disorders across five domains: physical signs and symptoms, sports, work, manner of living, and feelings. It ranges from 0 to 2100, and the lower the total, the better the result.
Inclinometer | 5-6weeks
  The inclinometer calculates shoulder R.O.M. in degrees with high accuracy. These are flexion: 170-180° rotation, abduction: 170-180°, external rotation: 90°, and internal rotation: 70-90°.
Push-Up Plus Test | 5-6weeks
  The Push-Up Plus Test is designed to assess both scapular stability and serratus anterior muscle strength from the observed scapular movements during the 'plus' action in a push-up formation. They are either pass/fail scores or quantitative repet

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Islam, DPT, Principal Investigator — Riphah International University
Locations (1):
- Combined Military Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abufoul R, Gavish L, Haddad M. Photobiomodulation self-treatment at home after rotator cuff arthroscopic repair accelerates improvement in pain, functionality, and quality of life: A double-blind, sham-controlled, randomized clinical trial. Lasers Surg Med. 2023 Sep;55(7):662-673. doi: 10.1002/lsm.23692. Epub 2023 Jun 8. PMID 37288499
- [Background] Cools AM, Maenhout AG, Vanderstukken F, Decleve P, Johansson FR, Borms D. The challenge of the sporting shoulder: From injury prevention through sport-specific rehabilitation toward return to play. Ann Phys Rehabil Med. 2021 Jul;64(4):101384. doi: 10.1016/j.rehab.2020.03.009. Epub 2020 Apr 29. PMID 32320753
- [Background] AlAnazi A, Alghadir AH, Gabr SA. Handgrip Strength Exercises Modulate Shoulder Pain, Function, and Strength of Rotator Cuff Muscles of Patients with Primary Subacromial Impingement Syndrome. Biomed Res Int. 2022 Aug 30;2022:9151831. doi: 10.1155/2022/9151831. eCollection 2022. PMID 36082154
- [Background] Kesikburun S, Tan AK, Yilmaz B, Yasar E, Yazicioglu K. Platelet-rich plasma injections in the treatment of chronic rotator cuff tendinopathy: a randomized controlled trial with 1-year follow-up. Am J Sports Med. 2013 Nov;41(11):2609-16. doi: 10.1177/0363546513496542. Epub 2013 Jul 26. PMID 23893418
- [Background] Camargo PR, Alburquerque-Sendin F, Salvini TF. Eccentric training as a new approach for rotator cuff tendinopathy: Review and perspectives. World J Orthop. 2014 Nov 18;5(5):634-44. doi: 10.5312/wjo.v5.i5.634. eCollection 2014 Nov 18. PMID 25405092
- [Background] Schedler S, Brueckner D, Hagen M, Muehlbauer T. Effects of a Traditional versus an Alternative Strengthening Exercise Program on Shoulder Pain, Function and Physical Performance in Individuals with Subacromial Shoulder Pain: A Randomized Controlled Trial. Sports (Basel). 2020 Apr 13;8(4):48. doi: 10.3390/sports8040048. PMID 32294940
- [Background] Bourke J, Skouteris H, Hatzikiriakidis K, Fahey D, Malliaras P. Use of Behavior Change Techniques Alongside Exercise in the Management of Rotator Cuff-Related Shoulder Pain: A Scoping Review. Phys Ther. 2022 Apr 1;102(4):pzab290. doi: 10.1093/ptj/pzab290. PMID 34972867
- [Background] Jones BH, Canham-Chervak M, Sleet DA. An evidence-based public health approach to injury priorities and prevention recommendations for the u.s. Military. Am J Prev Med. 2010 Jan;38(1 Suppl):S1-10. doi: 10.1016/j.amepre.2009.10.001. PMID 20117582
- [Background] Jones A, Sealey R, Crowe M, Gordon S. Concurrent validity and reliability of the Simple Goniometer iPhone app compared with the Universal Goniometer. Physiother Theory Pract. 2014 Oct;30(7):512-6. doi: 10.3109/09593985.2014.900835. Epub 2014 Mar 25. PMID 24666408
- [Background] Keene DJ, Soutakbar H, Hopewell S, Heine P, Jaggi A, Littlewood C, Hansen Z, Barker K, Hamilton W, Carr AJ, Lamb SE. Development and implementation of the physiotherapy-led exercise interventions for the treatment of rotator cuff disorders for the 'Getting it Right: Addressing Shoulder Pain' (GRASP) trial. Physiotherapy. 2020 Jun;107:252-266. doi: 10.1016/j.physio.2019.07.002. Epub 2019 Jul 9. PMID 32026827